CLINICAL TRIAL: NCT01805297
Title: Intravitreal Aflibercept Injection as a Surgical Adjuvant in Severe Proliferative Diabetic Retinopathy
Brief Title: Aflibercept Injection for Proliferative Diabetic Retinopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2148
Record Dates: First submitted 2013-02-26; First posted 2013-03-06 (Estimated); Results first posted 2017-09-13 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Vitreous Hemorrhage
Keywords: Proliferative Diabetic Retinopathy
MeSH Terms: conditions — Vitreous Hemorrhage | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitrectomy with Aflibercept Injection (Active Comparator): Preoperative 2.0mg intravitreal aflibercept and vitrectomy with intraoperative 2.0mg intravitreal aflibercept injection.
  Interventions: Drug: Intravitreal Aflibercept Injection
- Standard Vitrectomy (Active Comparator): Preoperative 2.0mg intravitreal aflibercept and standard of care vitrectomy.
  Interventions: Other: Standard Vitrectomy

INTERVENTIONS:
Drug: Intravitreal Aflibercept Injection — One time 2.0mg aflibercept injection, following pars plana vitrectomy.
  Other Names: Eylea
  Arms: Vitrectomy with Aflibercept Injection
Other: Standard Vitrectomy — Surgical intervention
  Arms: Standard Vitrectomy

SUMMARY:
To evaluate the ocular and systemic safety of intravitreal aflibercept injection in patients undergoing Pars Plana Vitrectomy for Proliferative Diabetic Retinopathy.

DETAILED DESCRIPTION:
Patients who need Pars Plana Vitrectomy surgery, and agree to participate in this study will receive an injection of 2.0mg aflibercept 4 to 6 days before Vitrectomy surgery. Half of these patients will be randomized to receive another injection of 2.0mg aflibercept immediately after their surgery. Postoperative patient visits in this study will be at 1 day, and at weeks 1, 4, 16 and 24, and at any other times as deemed necessary by the Investigator.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 18 years
* Diagnosed with proliferative diabetic retinopathy (PDR) requiring pars plana vitrectomy (PPV)
* Best corrected visual acuity in the study eye between 20/40 to light perception (LP) using an Early Treatment Diabetic Retinopathy Study (ETDRS) chart

Exclusion Criteria:

* Pregnancy (positive urine pregnancy test) or lactation
* Premenopausal women not using adequate contraception. The following are considered effective means of contraception: surgical sterilization or use of oral contraceptives, barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel, an intrauterine device (IUD), or contraceptive hormone implant or patch.
* Participation in a study of an investigational drug or device within the past 30 days prior to enrolling in the study
* For previously treated subjects -
* Prior treatment with anti-vascular endothelial growth factor (anti-VEGF) therapy in the study eye within 28 days of Screening
* Prior treatment with triamcinolone in the study eye within 6 months of Screening.
* Prior treatment with dexamethasone in the study eye within 30 days of Screening
* Intraocular surgery (including cataract surgery) in the study eye within 2 months preceding Baseline
* History of vitrectomy surgery, submacular surgery, or other surgical intervention for PDR in the study eye
* Active intraocular inflammation (grade trace or above) in the study eye
* History of rhegmatogenous retinal detachment or macular hole (Stage 3 or 4) in the study eye
* Active infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye
* Uncontrolled glaucoma in the study eye (defined as intraocular pressure (IOP) ≥ 30 mmHg despite treatment with anti-glaucoma medication)
* History of cerebral vascular accident, myocardial infarction, transient ischemic attacks within 6 months of study enrollment.
* History of allergy to fluorescein, indocyanine green (ICG) or iodine, not amenable to treatment
* Presence of macular traction
* Uncontrolled hypertension (e.g., 120/200 mmHg) prior to surgery (PPV)
* Concomitant use of any systemic anti-VEGF therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-03; Primary Completion 2014-02 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert E Leonard, MD, Principal Investigator — Dean McGee Eye Institute; Vinay A Shah, MD, Principal Investigator — Dean McGee Eye Institute
Locations (1):
- Dean McGee Eye Institute, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dervenis P, Dervenis N, Smith JM, Steel DH. Anti-vascular endothelial growth factors in combination with vitrectomy for complications of proliferative diabetic retinopathy. Cochrane Database Syst Rev. 2023 May 31;5(5):CD008214. doi: 10.1002/14651858.CD008214.pub4. PMID 37260074

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vitrectomy With Aflibercept Injection | Standard Vitrectomy
Started | 6 | 6
Completed | 4 | 3
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Vitrectomy With Aflibercept Injection: Preoperative 2.0mg intravitreal aflibercept and vitrectomy with intraoperative 2.0mg intravitreal aflibercept injection.
  Intravitreal Aflibercept Injection: One time 2.0mg aflibercept injection, immediately following pars plana vitrectomy.
- Total: Total of all reporting groups
Arm/Group | Vitrectomy With Aflibercept Injection | Standard Vitrectomy | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 11
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 3 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 4 | 5 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12
Mean visual acuity [Mean (Full Range); unit: number of letters read on ETDRS Chart] — Number of letters read on the "Early Treatment Diabetic Retinopathy Study" visual acuity chart. a higher number indicates a better visual acuity (example, 0 means no letters could be read while 100 means all 100 letters present on chart were read)
  number of letters read on ETDRS Chart | 13.8 [0 to 100] | 17.7 [0 to 100] | 15.9 [0 to 100]
Intraocular pressure [Mean (Full Range); unit: mmHg] | 14 [10 to 18] | 11.2 [6 to 18] | 12.6 [6 to 18]
Central retinal thickness [Mean (Full Range); unit: Microns] — Population: Optical Coherence Tomography performed only as visualization permitted
  Microns
    number analyzed (Participants) | 1 | 1 | 2
    (all) | 304 [304 to 304] | 305 [305 to 305] | 304.5 [304 to 305]

OUTCOME MEASURES:

1. Primary Outcome: Rate of Resolved Post-operative Vitreous Hemorrhage.
Description: Percentage of patients who had no vitreous hemorrhage before or at week 24
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Vitrectomy With Aflibercept Injection | Standard Vitrectomy
Number analyzed (Participants) | 6 | 6
Participants | 6 | 5

2. Secondary Outcome: Mean Change in Visual Acuity
Description: Change in visual acuity measured using "Early Treatment of Diabetic Retinopathy Study" visual acuity charts and letter score difference from baseline to 6 month. A greater number indicates a higher increase in vision from the baseline score. A negative number would indicate that vision decreased.
Time Frame: 24 weeks
Population: Patients who completed 24 week visit
Measure: Mean (Full Range); unit: Number of letters Read
Arm/Group | Vitrectomy With Aflibercept Injection | Standard Vitrectomy
Number analyzed (Participants) | 4 | 3
Number of letters Read | 56.75 [0 to 100] | 41.67 [0 to 100]

3. Secondary Outcome: Need for Any Additional Surgical Intervention.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Vitrectomy With Aflibercept Injection | Standard Vitrectomy
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

4. Secondary Outcome: Changes in Mean Central Retinal Thickness.
Description: The amount of thickness change in microns from baseline to 6 month visit. A positive number indicates an increase in thickness and a negative number would indicate a decrease in thickness.
Time Frame: 24 weeks
Population: Due to lack of clear view due to vitreous Hemorrhage, all but 2 patients were unable to have optical coherence tomography at baseline, and one these was lost to follow up. For this reason, data collected for the few patients who were able to have the test was not analyzed
Measure: Number; unit: Microns
Arm/Group | Vitrectomy With Aflibercept Injection | Standard Vitrectomy
Number analyzed (Participants) | 0 | 1
Microns |  | 20

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Vitrectomy With Aflibercept Injection | Standard Vitrectomy
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 6/6 | 5/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitrectomy With Aflibercept Injection (N=6) | Standard Vitrectomy (N=6)
Headache (General disorders) | 1 (1) | 3 (3)
Broken Rib (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Post operative ocular pain (Eye disorders) | 3 (3) | 4 (4) — pain after vitrectomy surgery
descemet's folds (Eye disorders) | 0 (0) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Subconjunctival Hemorrhage (Eye disorders) | 2 (2) | 1 (1) — sub conjunctival hemorrhage occurring post treatment
vitreous haze (Eye disorders) | 1 (1) | 0 (0) — vitreous haze occurring in non-study eye
cataract (Eye disorders) | 0 (0) | 1 (1) — worsening of cataract post operatively
Optic disc pallor (Eye disorders) | 0 (0) | 1 (1) — observed on clinical exam
visual disturbance (Eye disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) — post operative nausea
vitreous hemorrhage (Eye disorders) | 1 (1) | 0 (0) — seen in non study eye on clinical exam
photophobia (Eye disorders) | 1 (1) | 0 (0)
tooth decay (General disorders) | 1 (1) | 1 (1)
tongue injury (General disorders) | 1 (1) | 0 (0) — patient reported biting and injuring tongue
ocular irritation (Eye disorders) | 0 (0) | 1 (1) — patient reported ocular irritation post operatively

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No